CLINICAL TRIAL: NCT04363632
Title: Prospective Analysis of Morbi-mortality of Patients With Cancers in Active Phase of Treatment Suspected or Diagnosed of a SARS-CoV-2 Infection
Acronym: ONCOVID-19
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET20-069
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Sars-CoV2; Cancer
Keywords: COVID-19; Oncology; Epidemiology; Predictive factors
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
National multicentre epidemiological study to describe retrospectively and prospectively the clinical outcomes of patients with a suspected coronavirus infection (either confirmed or not) while receiving a medical treatment for the underlying cancer

ELIGIBILITY:
Inclusion Criteria:

I1. Confirmed diagnosis of any type of solid or hematologic tumor;

I2. Ongoing anticancer treatment (cytotoxic, targeted therapy, immunotherapy or loco regional procedure, including radiotherapy, surgery or interventional radiology procedure) at the time of inclusion or within the last 3 months prior to inclusion (last treatment administration or last loco regional procedure) ;

I3. Patient with suspicion of COVID-19 (clinical symptoms of COVID-19 including fever (>38°C) and/or respiratory tract symptoms), either confirmed or not.

Note 1: Patients must have underwent diagnostic procedures: diagnostic test (positive or negative) and/or chest imaging. Note 2: Patients will be eligible regardless of the presence of a neutropenia (either febrile or not) ;

I4. Patient and/or family did not decline data collection after complete information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cancer in active phase of treatment suspected or diagnosed of a SARS-CoV-2 infection
Sampling Method: Probability Sample
Enrollment: 1231 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Mortality of cancer patients under active anticancer treatment | 28 days after the date of the diagnostic procedure
  Mortality rate, defined as the proportion of patients who are dead 28 days after the date of the diagnostic procedure for the 2 cohorts of patients (positive and negative).

SECONDARY OUTCOMES:
Overall survival | 6 months (i.e. at the the time of last patient last visit)
  Overall survival will be defined as the time from the date of the first diagnostic procedure (either diagnostic test or chest imaging) to the date of death due to any cause.
Hospitalizations | 28 days after the date of the diagnostic procedure
  The duration of hospitalization (from the date of hospitalization to the date of definitive discharge for live patients)
Death | 6 months (i.e. at the the time of last patient last visit)
  Cause of death, related or not to the COVID-19
Complications | 28 days after the date of the diagnostic procedure
  Associated complications described by their type
Hospitalizations | 28 days after the date of the diagnostic procedure
  proportion of hospitalizations
Patients' characteristics | At the date of the diagnostic procedure
  To describe accurately patients' characteristics in terms of demographics
Patients' characteristics | At the date of the diagnostic procedure
  To describe accurately patients' characteristics in type of tumor
Patients' characteristics | At the date of the diagnostic procedure
  To describe accurately patients' characteristics in type of anticancer treatment,
Patients' characteristics | At the date of the diagnostic procedure
  To describe accurately patients' characteristics in terms of comorbidities

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Hospitalier Métropole Savoie, Chambéry
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - CH Annecy-Genevois, Metz-Tessy
  - Groupement Hospitalier Porte de Provence, Montélimar
  - Institut de Cancérologie de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg
  - Institut Universitaire du Cancer de Toulouse - IUCT Oncopole, Toulouse
  - CH Valence, Valence

REFERENCES:
- [Derived] Assaad S, Zrounba P, Cropet C; ONCOVID-19 study Consortium; Blay JY. Mortality of patients with solid and haematological cancers presenting with symptoms of COVID-19 with vs without detectable SARS-COV-2: a French nationwide prospective cohort study. Br J Cancer. 2021 Aug;125(5):658-671. doi: 10.1038/s41416-021-01452-4. Epub 2021 Jun 16. PMID 34135471